CLINICAL TRIAL: NCT03911635
Title: Applying of Urethral Advancement, Glanuloplasty and Preputioplasty Technique for More Proximal Degrees of Hypospadias. Selective Criteria and a Modified Technique
Brief Title: Selective Criteria and a Modified Technique of Applying "URAGPI" Technique for More Proximal Degree of Hypospadias
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ali Ahmed, Principal Investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: URAGPI in hypospadias
Record Dates: First submitted 2019-03-23; First posted 2019-04-11 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Hypospadias
MeSH Terms: conditions — Hypospadias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hypospadias in children (Experimental): Distal shaft hypospadias at age of 12 years or less
  Interventions: Procedure: URAGPI technique

INTERVENTIONS:
Procedure: URAGPI technique — the Urethral Advancement, Glanuloplasty and Preputioplasty

SUMMARY:
Hypospadias is a condition in which the location of the urethral meatus is on the ventral aspect of the penis.

Hypospadias is the most common congenital anomaly of urogenital organs in boys, with an incidence of approximately 1 in 250 newborns. Recently, case selection has been advised to avoid possible complications and limitations [1]. The meatal advancement and glanuloplasty (MAGPI) procedure was first described in 1981 for the repair of distal hypospadias. An excellent surgical result requires careful case selection, avoiding cases with thin or rigid ventral para-meatal skin or a meatus too proximal or too wide. The glans wrap to support the advanced ventral urethral wall requires a solid tissue approximation in two layers to prevent regression of the meatus. Meatal stenosis can be avoided by assuring an adequate dorsal Heineke- Mikulicz tissue rearrangement and making an incision from within the urethral meatus well distally into the urethral groove. . The overall success rate with the MAGPI procedure suggests that it should continue to be used in the repair of distal hypospadias [2]. The advantage of Urethral advancement, Glanuloplasty, and Preputioplasty " URAGPI" versus MAGPI Is that A) Applicability to almost any type of distal hypospadias regardless of the severity of glanular ventriflexion.

B) Normal appearance of the penis. C) Good functional results.

ELIGIBILITY:
Inclusion Criteria:

* All patient with hypospadias from 1 to 12 years with penile selection according to Wang YN et. al

Exclusion Criteria:

* circumcised patients
* sever degrees of chordae
* previous surgical repair
* meatal stenosis

Ages: 1 Year to 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75 (Estimated)
Dates: Start 2020-04-01 (Estimated); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of the patient immediately after removal of the catheter at the 7th day and after 3 weeks | 3 weeks
  evaluation according to "Hypospadias Objective Penile Evaluation Score"